CLINICAL TRIAL: NCT01686971
Title: The Needs of Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0044-12rmb.ctil
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Needs and Demands of Oncology Patients; Breast Cancer Patients.; Colon Cancer Patients.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- questionaire: patients will receive a questionaire and speak to a nurse regarding their needs and/ or demands.

SUMMARY:
A questionaire for cancer patients without an active treatment in order to evaluate their needs and/or demands.

DETAILED DESCRIPTION:
Cancer patients on finishing therapy will be interviewed by a registered nurse by a approved questionaire asking about his /her feeling needs and demands.

Efforts to help them will be trid

It is well known from studies that survivors have unmet medical and non-medical needs that are not met, this includes physical, emotional and practical issues. The purpose of this study is to study them and investigate the methods how to alleviate them.

All patients with breast and colon cancer that are refered to the Rambam Oncology center will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with two common cancers (breast, colon) that have completed the treatment (chemotherapy, radiotherapy)
* Male and Female patients 18-80 years old.

Exclusion Criteria:

* Patients with active disease.
* Recipients of care that matches the criteria of hospice care.
* Patients with a diagnosis of dementia or other cognitive failure
* Patients who do not speak Hebrew

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology patients at the end of theier treatment. The patients will consist from 2 most common cancer diseases:Breast cancer and colon cancer.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-05 (Estimated); Study Completion 2013-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eliezer Robinson, Proffesor, Principal Investigator — Rambam MC
Locations (1):
- Rambam MC, Haifa, Israel